CLINICAL TRIAL: NCT03460678
Title: Randomized Multicenter Study to Compare the Effectiveness and Safety of Erlotinib and Pemetrexed as Maintenance Therapy of Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Randomized Comparative Study of Erlotinib and Pemetrexed in the Maintenance Treatment of Advanced Lung Cancer Patients.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRT-JOR-LEB-KSA-2016-04
Record Dates: First submitted 2018-02-26; First posted 2018-03-09 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Generic Erlotinib; Generic Pemetrexed; NSCLC; Non-squamous; Randomized Study; Maintenance Therapy; Tyrosine kinase inhibitor; Antifolate antineoplastic agents
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized into either the arm of Erlotinib 150 mg once daily, or the arm of Pemetrexed 500 mg/m2 administered as an intravenous infusion over 10 minutes on the first day of each 21-day cycle, until disease progression or unacceptable toxic effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pemetrexed Arm (Other): Vials containing powder for concentrate for solution for infusion equivalent to 500 mg of pemetrexed (as disodium)
  Interventions: Drug: Pemetrexed
- Erlotinib Arm (Other): Film coated tablets containing 150 mg erlotinib (as erlotinib hydrochloride)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Pemetrexed — Vials containing powder for concentrate for solution for infusion equivalent to 500 mg of pemetrexed (as disodium) administered as 500mg/m2 IV over 10 minutes on the first day of each 21-day cycle, until disease progression or unacceptable toxic effects
  Other Names: Pemitra®
  Arms: Pemetrexed Arm
Drug: Erlotinib — Film coated tablets containing 150 mg erlotinib (as erlotinib hydrochloride) administered once daily until disease progression or unacceptable toxic effects
  Other Names: Mirata®
  Arms: Erlotinib Arm

SUMMARY:
The purpose of this multicenter randomized study is to compare the effectiveness and safety of erlotinib and pemetrexed in the maintenance treatment of patients with advanced non-squamous non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
A randomized multi-center prospective study to compare the 12-month effectiveness (survival) and safety of erlotinib and pemetrexed as maintenance treatment in two groups of patients with locally advanced or metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC) other than predominantly squamous cell histology, whose disease has not progressed immediately following platinum-based chemotherapy for 4 cycles administered per routine daily practice in each study center

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Signed written informed consent
* Histologically or cytological diagnosed stage IIIB/IV non-squamous histology NSCLC
* Received platinum based doublet chemotherapy for 4 cycles as first line therapy before this study
* Patients upon enrolment has at least stable disease following the platinum doublet; with documented (confirmed or unconfirmed) radiographic evidence of a tumor response of complete response (CR), partial response (PR), or stable disease (SD) according to RECIST version 1.1 criteria
* Estimated Life expectancy ≥ 3 months
* Eastern cooperative oncology group performance status (ECOG PS) 0-2
* Adequate organ function

Exclusion Criteria:

* Age ˂18 years
* Predominantly squamous cell and/or mixed small cell, non-small cell histology
* Current treatment on another therapeutic clinical study or within the last 30 days of entering the study
* Spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function, carcinomatous meningitis, or leptomeningeal disease
* Any of the following within the 3 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack
* Ongoing cardiac dysrhythmias of national cancer institute-common terminology criteria for adverse events (NCI CTCAE) Grade >2, uncontrolled atrial fibrillation of any grade, or corrected QT interval (QTc) >470 msec
* Pregnancy or breastfeeding
* Prior malignancy (other than current NSCLC): patients will not be eligible if they have evidence of active malignancy (other than non-melanoma skin cancer or localized cervical cancer, or localized and presumed cured prostate cancer) within the last 3 years
* Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities that would impose, in the judgment of the investigator and/or sponsor, excessive risk associated with study participation or study drug administration, and which would, therefore, make the patient inappropriate to enter this study
* Uncontrolled third-space fluid collections
* Progressive brain metastases
* Hypersensitivity to the study drugs
* Inability to take corticosteroid drugs, folic acid, or vitamin B12
* Patients with epidermal growth factor receptor (EGFR) positive, anaplastic lymphoma kinase (ALK) positive (documented using fluorescence in situ hybridization (FISH) and/or immunohistochemistry (IHC)), or unknown EGFR and ALK test results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in eligible patients randomized to erlotinib or pemetrexed treatment arms | 12 months
  Progression Free Survival is defined as the time from date of randomization to the date of tumor progression or death from any cause, assessed until at least 12 months after randomization.
  Progression is defined using response evaluation criteria in solid tumors (RECIST version 1.1)

SECONDARY OUTCOMES:
Median Overall Survival (OS) Time between eligible patients randomized to erlotinib or pemetrexed treatment of therapy | 12 months
  Overall survival time is defined as the time from date of randomization until the date of death from any cause, assessed until at least 12 months after randomization
Overall response rate and duration between eligible patients randomized to erlotinib or pemetrexed treatment arms | 12 months
  Overall response defined using RECIST version 1.1 and the duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or progressive disease (PD) is objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started) or until at least 12 months after randomization as assessed every 6 weeks
Incidence of adverse events (AEs) and serious adverse events (SAEs) to erlotinib and pemetrexed | 12 months
  Incidence rates, severity, relationship of adverse events (AEs) and serious AE (SAE) to treatment drugs, number of AEs leading to permanent treatment discontinuation and clinically relevant changes in laboratory tests will be recorded, estimated and presented

CONTACTS AND LOCATIONS:
Locations (2):
- King Hussein Cancer Center (KHCC), Amman, Jordan
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No